CLINICAL TRIAL: NCT06574464
Title: Predicting Mortality in Adults Hospitalized With Multiple Trauma: Can the BIG Score Estimate Risk?
Brief Title: The BIG Score and In-Hospital Trauma Mortality
Acronym: BIGstd
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Adem Az, Principal Investigator, Haseki Training and Research Hospital
Other Study IDs: 2023-202
Record Dates: First submitted 2024-08-25; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Multiple Trauma; Injury Traumatic
Keywords: BIG score; revised trauma score; injury severity score; mortality; multiple trauma
MeSH Terms: conditions — Multiple Trauma; Wounds and Injuries | interventions — Glasgow Coma Scale; Injury Severity Score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors: Survivors were defined as patients who were still alive after 28 days of admission to the emergency department.
  Interventions: Other: BIG SCORE; Other: Glasgow coma scale; Other: Revised Trauma Score; Other: Injury Severity Score
- Non-survivors: Non-survivors had passed away within 28 days of admission to the emergency department
  Interventions: Other: BIG SCORE; Other: Glasgow coma scale; Other: Revised Trauma Score; Other: Injury Severity Score

INTERVENTIONS:
Other: BIG SCORE — The trauma BIG score is used to predict posttraumatic injury severity and mortality. It was originally designed for the pediatric population. The score is calculated using the Base Deficit (BD), International Normalized Ratio (INR), and Glasgow Coma Scale (GCS) score on admission using the following formula:
  BIG score = (admission BD) + (2.5 × INR) + (15 - GCS).
Other: Glasgow coma scale — The Glasgow Coma Scale is a neurological assessment tool used to evaluate the level of consciousness of a patient. It assesses three items: eye-opening (spontaneous, 4 points; to verbal stimuli, 3 points; to pain stimuli, 2 points; no response, 1 point); verbal responses (oriented, 5 points; confused but coherent speech, 4 points; inappropriate words, 3 points; incomprehensible speech, 2 points; no response, 1 point); and motor responses (obeys commands, 6 points; localizes pain, 5 points; withdraws from pain, 4 points; flexes in response to pain, 3 points; extends in response to pain, 2 points; no response, 1 point). The total GCS score is obtained by summing the scores for the three items, and it ranges from 3 to 15.
Other: Revised Trauma Score — The Revised Trauma Score (RTS) is a physiological scoring system used to assess the severity of a traumatic injury. It considers three key parameters, Glasgow Coma Scale (GCS), Systolic Blood Pressure (SBP), and Respiratory Rate (RR), with a total score of 12 points. The study team retrospectively computed the RTS on admission by retrieving the GCS score, SBP, and RR per minute from the hospital's automated systems and archives.
Other: Injury Severity Score — The Injury Severity Score (ISS) is an anatomical scoring system used to assess the severity of injuries sustained by trauma patients. It provides a numerical value based on the anatomical regions of the body affected by trauma and the severity of those injuries. The ISS is calculated by dividing the body into six regions: the head/neck, face, chest, abdomen/pelvis, extremities, and external. Each region is assigned a score ranging from 1 to 6, with 1 indicating minor injury and 6 indicating severe injury. The highest score from each region is squared and then the scores are summed to calculate the overall ISS.

SUMMARY:
This study investigated the efficacy and reliability of the BIG score, calculated based on the base deficit (BD), International Normalized Ratio (INR), and Glasgow coma scale (GCS), in comparison with the GCS, Revised trauma score (RTS), and Injury Severity Score (ISS) for predicting in-hospital mortality in adults with multiple-trauma presenting to the emergency department (ED).

DETAILED DESCRIPTION:
This retrospective, observational, single-center study included 563 consecutive adults (≥ 18 years old) with multiple trauma who were admitted to our emergency department and hospitalized between January 2022 and December 2023. We assessed patient demographics (age and sex), vital signs on admission (systolic blood pressure [SBP, mmHg], heart rate [HR, beats/min], respiratory rate [RR, breaths/min], and peripheral oxygen saturation [SpO2, %]), complaints and symptoms on admission, anatomic region of injury, type of trauma (blunt or penetrating), mechanism of injury, BD measured in blood gases, INR, trauma scoring systems (e.g., GCS, RTS, ISS, and BIG score), and clinical outcomes (discharge, hospitalization, or death). The study cohort was divided into survivors and non-survivors. Survivors were defined as patients who were still alive after 28 days, while non-survivors had passed away within that time. The demographics, clinical characteristics, and trauma scoring systems were compared between survivors and non-survivors to determine the prognosis of patients with multiple trauma. Independent predictors of mortality were determined by multivariate logistic regression analysis of variables (demographic characteristics, clinical characteristics, and trauma scores) that differed significantly between survivors and non-survivors. Receiver operating characteristic (ROC) curve analysis was performed to establish cut-off values for the GCS, RTS, ISS, and BIG score, and then to assess the sensitivity and specificity of these scoring systems in terms of predicting in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* This study included 563 consecutive adults (≥ 18 years old) with multiple trauma who were admitted to our Emergency Department and hospitalized between January 2022 and December 2023.

Exclusion Criteria:

* Patients aged < 18 years and adults who were discharged from the Emergency Department
* Patients with non-traumatic injuries and those who presented to the Emergency Department for reasons other than trauma
* Patients with missing Base Deficit and International Normalized Ratio levels
* Patients who had been admitted to the hospital more than 24 hours after the trauma
* Patients with single trauma (e.g., isolated extremity trauma, isolated head injury, etc.)
* Patients with chronic conditions such as chronic renal failure or hepatic, hematological, or neurological diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective, observational, single-center study included 563 consecutive adults (≥ 18 years old) with multiple trauma who were admitted to our Emergency Department and hospitalized between January 2022 and December 2023. Our
Sampling Method: Probability Sample
Enrollment: 563 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Predictive ability of BIG score for 28-day mortality | From admission to 28 days
  The investigators assessed the predictive ability of BIG score in determining 28-day mortality.
Predictive ability of Glasgow coma scale for 28-day mortality | From admission to 28 days
  The investigators assessed the predictive ability of Glasgow coma scale in determining 28-day mortality.
Predictive ability of Revised Trauma Score for 28-day mortality | From admission to 28 days
  The investigators assessed the predictive ability of Revised Trauma score in determining 28-day mortality.
Predictive ability of Injury Severity Score for 28-day mortality | From admission to 28 days
  The investigators assessed the predictive ability of Injury Severity Score in determining 28-day mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Adem Az, M.D., Principal Investigator — Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Stored in non-publicly available Available on request

REFERENCES:
- [Result] Hoke MH, Usul E, Ozkan S. Comparison of Trauma Severity Scores (ISS, NISS, RTS, BIG Score, and TRISS) in Multiple Trauma Patients. J Trauma Nurs. 2021 Apr-Jun 01;28(2):100-106. doi: 10.1097/JTN.0000000000000567. PMID 33667204
- [Result] Borgman MA, Maegele M, Wade CE, Blackbourne LH, Spinella PC. Pediatric trauma BIG score: predicting mortality in children after military and civilian trauma. Pediatrics. 2011 Apr;127(4):e892-7. doi: 10.1542/peds.2010-2439. Epub 2011 Mar 21. PMID 21422095
- [Result] Brockamp T, Maegele M, Gaarder C, Goslings JC, Cohen MJ, Lefering R, Joosse P, Naess PA, Skaga NO, Groat T, Eaglestone S, Borgman MA, Spinella PC, Schreiber MA, Brohi K. Comparison of the predictive performance of the BIG, TRISS, and PS09 score in an adult trauma population derived from multiple international trauma registries. Crit Care. 2013 Jul 11;17(4):R134. doi: 10.1186/cc12813. PMID 23844754
- [Result] Park S, Wang IJ, Yeom SR, Park SW, Cho SJ, Yang WT, Tae W, Huh U, Song C, Kim Y, Park JH, Cho Y. Usefulness of the BIG Score in Predicting Massive Transfusion and In-Hospital Death in Adult Trauma Patients. Emerg Med Int. 2023 Oct 17;2023:5162050. doi: 10.1155/2023/5162050. eCollection 2023. PMID 37881258
- [Derived] Az A, Sogut O, Ozcomlekci M, Dogan Y, Akdemir T. Predicting mortality in adults hospitalized with multiple trauma: Can the BIG score estimate risk? Ulus Travma Acil Cerrahi Derg. 2025 Jan;31(1):66-74. doi: 10.14744/tjtes.2024.92879. PMID 39775514